CLINICAL TRIAL: NCT01081548
Title: A Multi-center, Randomized, Open-labeled Clinical Trial to Evaluate Efficacy and Safety of Lipinon® 20mg Versus Lipitor® 20mg in Korean Patients With Hypercholesterolemia
Brief Title: A Clinical Trial Study to Evaluate Efficacy and Safety of Atorvastatin in Korean Patients With Hypercholesterolemia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Dong Hoon Choi/Prof., Dept of Cardiology/Severance Hospital/Yonsei U
Model: Parallel | Masking: None
Other Study IDs: 4-2008-0288
Record Dates: First submitted 2010-03-04; First posted 2010-03-05 (Estimated); Last update posted 2010-03-05 (Estimated); Status verified 2010-01

CONDITIONS: Hypercholesterolemia
MeSH Terms: conditions — Hypercholesterolemia | interventions — Atorvastatin

ARMS (2):
- Generic (Experimental)
  Interventions: Drug: atorvastatin
- Lipitor (Active Comparator)
  Interventions: Drug: atorvastatin

INTERVENTIONS:
Drug: atorvastatin — 20 mg
  Other Names: Lipinon
  Arms: Generic
Drug: atorvastatin — 20 mg
  Other Names: Lipitor
  Arms: Lipitor

SUMMARY:
The purpose of this study is to compare the efficacy and safety of atorvastatin generic product with reference drug.

ELIGIBILITY:
Inclusion Criteria:

* Age 20 ~ 79
* People who have not reached LDL-C targeted level in accordance with the guidelines for hyperlipidemia management released by Korean Society of Lipidology and Atherosclerosis
* In case of female participants taking combination HRT or oral contraceptive, they should maintain stable capacity and usage at least for 8 weeks before the visit 1.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2008-08; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Severance Hospital, Seoul, South Korea